CLINICAL TRIAL: NCT05677087
Title: PREPARE Project: Examining Impacts of the COVID-19 Pandemic on Maternal Health and Infant and Young Child Feeding Practices
Brief Title: PREPARE: Remote Nutrition Education, Ghana
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Collaborators: University of Ghana (Other)
Responsible Party: Principal Investigator, Ruthfirst Ayande, Principal Investigator, University of Massachusetts, Amherst
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2578
Record Dates: First submitted 2022-12-14; First posted 2023-01-10 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Health Literacy; Dietary Diversity; Infant Feeding Practices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prepare project education (Experimental): This group will receive an intensive 6-week remote nutrition education intervention
  Interventions: Behavioral: PREPARE Nutrition Education Module

INTERVENTIONS:
Behavioral: PREPARE Nutrition Education Module — The Perinatal Remote Education for Pandemic Resilience (PREARE) program is a 6-week intensive program aimed at increasing maternal and infant dietary diversity as well as maternal health literacy. Modules that will be completed in the program include education on early initiation of breastfeeding, food groups and the benefits of a balanced diet, appropriate meal frequency for mother and infant, and appropriate sources of health information. Information on personal hygiene and COVID-19 hygiene protocols as well as danger signs during pregnancy are included in the module to improve maternal knowledge on safety protocols and pregnancy complications.

SUMMARY:
In the wake of the pandemic, it is important to explore remote nutrition education programs during the pre- and postnatal period. This is the second phase of a bigger project, where a 6-week intensive remotely delivered nutrition and health education program called the PREPARE program will be piloted. Prepare stands for "Perinatal Remote Education for Pandemic Resilience", and it is a nutrition and health education program meant for pregnant and lactating women aimed at improving maternal and infant dietary diversity, maternal health literacy and increasing COVID-19 awareness. One hundred women will be selected from a pool of 233 women who completed a baseline survey last year. Fifty of them will receive the intervention and the other 50 will receive a delayed intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women currently enrolled on the preliminary phase of the PREPARE project who participated in our baseline survey are eligible. To have been part of the preliminary survey, women had to have had children between 6 and 15 months old during recruitment last year.
* Due to our primary outcome of infant dietary diversity, women from our preliminary survey whose children are currently between 6 months and 2 years will be included in the PREPARE pilot study.

Exclusion Criteria:

* In our preliminary survey, participants were excluded if they were non-Ghanaian or currently pregnant.
* Besides women who had children less than 6 months at time of recruitment, there will be no other exclusion criteria for the PREPARE pilot.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Study focuses on women with children born during the pandemic
Enrollment: 65 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
% infants meeting the Minimum Dietary Diversity (MDD) | 6 weeks
  Dietary diversity refers to the number of food items consumed from WHO classified food groups over a reference period (FAO, 2016). To meet the minimum dietary diversity, infants should have consumed 4 out of 7 food groups based on a 24-hr dietary recall and the WHO food group classification: 1. grains, roots and tubers, 2. legumes and nuts, 3. dairy products (milk, yogurt, cheese), 4. flesh foods (meat, fish, poultry and liver/organ meats), 5. Eggs, 6. vitamin-A rich fruits and vegetables, 7. other fruits and vegetables
% of Mothers meeting the Minimum Dietary Diversity for women (MDD-W) | 6 weeks
  Number of food items consumed from WHO classified food groups over a reference period (FAO, 2016). To meet the minimum dietary diversity, mothers should have consumed 5 out of 10 food groups based on a 24-hr dietary recall and the WHO food group classification: 1. Grains, white roots and tubers, and plantains, 2. Pulses (beans, peas and lentils) 3. Nuts and seeds 4. Dairy 5. Meat, poultry and fish 6. Eggs 7. Dark green leafy vegetables 8. Other vitamin A-rich fruits and vegetables 9. Other vegetables 10. Other fruits
% of mothers scoring >66% on the maternal health literacy inventory in pregnancy (MHELIP) scale. | 6 weeks
  Maternal health literacy (MHL) is the cognitive and social skills which determine the motivation and ability of individuals (mothers) to gain access to, understand and use information in ways which maintain and promote health for they and their children (Renkert and Nutbeam, 2001). This will be measured on the maternal health literacy inventory in pregnancy (MHELIP) scale (Taheri et al., 2020).

CONTACTS AND LOCATIONS:
Overall Officials: Ruthfirst EA Ayande, MSc, Principal Investigator — University of Massachusetts, Amherst; Elena T Carbone, DrPH, Study Chair — University of Massachusetts, Amherst
Locations (1):
- University of Ghana, Accra, Ghana